CLINICAL TRIAL: NCT04073823
Title: A Feasibility Study Evaluating Flexitouch® Plus With a Therapy Cycle Software Modification in Patients With Unilateral Breast Cancer-Related Lymphedema (BCRL)
Brief Title: A Study Evaluating FT-SW in Unilateral Breast Cancer-Related Lymphedema Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to unforeseen slow enrollment and a shift in corporate resources due to the COVID-19 impact.
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4070
Record Dates: First submitted 2019-07-25; First posted 2019-08-29 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer Related Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Flexitouch Plus (Active Comparator)
  Interventions: Device: Flexitouch Plus
- Flexitouch Plus with SW (Experimental)
  Interventions: Device: Flexitouch Plus FT with software modification

INTERVENTIONS:
Device: Flexitouch Plus — Flexitouch Plus full arm and core treatment
  Arms: Flexitouch Plus
Device: Flexitouch Plus FT with software modification — Flexitouch Plus full arm and trunk/chest treatment
  Other Names: FT-SW
  Arms: Flexitouch Plus with SW

SUMMARY:
The objective of the study is to demonstrate equivalency in treatment effect, as determined by objective measurements, between the modified therapy cycle software and the FDA-cleared Flexitouch therapy cycle software.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years of age or older
* Diagnosis of unilateral breast cancer-related lymphedema
* Stage I or early stage II lymphedema without severe fibrosis at the time of enrollment
* ≥ 5% volume difference between affected and unaffected arm as verified via perometry
* Willing and able to give informed consent
* Willing and able to comply with the study protocol requirements and all study-related visit requirements

Exclusion Criteria:

* In-home use of PCD within previous 3 months
* Therapist or self-administered manual lymph drainage (MLD) within previous 1 week
* Mastectomy or lymph node removal on side without lymphedema
* Bilateral lymphedema
* Heart failure (acute pulmonary edema, decompensated acute heart failure)
* Acute venous disease (acute thrombophlebitis, acute deep venous thrombosis, acute pulmonary embolism)
* Active skin or limb infection/inflammatory disease (acute cellulitis, other uncontrolled skin or untreated inflammatory skin disease) on the arms or trunk
* Active cancer (cancer that is currently under treatment, but not yet in remission)
* Poorly controlled kidney disease (glomerular filtration rate < 30 mls per minute), hypoproteinemia, pulmonary hypertension, hypothyroidism, cyclic edema, or Munchausen Syndrome
* BMI >50
* Any circumstance where increased lymphatic or venous return is undesirable
* Currently pregnant or trying to become pregnant
* Allergy to iodine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 53 [53 to 53] | 81 [81 to 81] | 67 [53 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Lymphatic Activation
Description: Comparison of the change in the rate of lymphatic propulsion events from the pre-treatment values to the post-treatment values for both the affected and contralateral limbs using the investigational technique of near infrared-fluorescent (NIRF) imaging.
Time Frame: Baseline and following a single treatment, an average of one hour
Measure: Number; unit: Percent Rate Change
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Percent Rate Change
  Affected Limb | 0.0 | -50
  Contralateral Limb | -3.0 | 241.2

2. Primary Outcome: Changes in Swelling - MoistureMeterD
Description: Comparison of the percent change in local tissue water from the pre-treatment values to the post-treatment values on the affected limb using MoistureMeterD.
Time Frame: Baseline and following a single treatment, an average of one hour
Measure: Mean (Full Range); unit: Percent Change
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Percent Change | -4.0 [-7.4 to 0.0] | -6.4 [-11.4 to 3.8]

3. Primary Outcome: Changes in Swelling - Perometry
Description: Swelling in the affected and contralateral limb as assessed using local tissue water content
Time Frame: Baseline and following a single treatment, an average of one hour
Measure: Number; unit: Percent Change
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Percent Change
  Affected Limb | 1.6 | -1.6
  Contralateral Limb | 0.5 | 0.7

4. Primary Outcome: Percent Change in Skin Thickness From Baseline to After Treatment.
Description: Skin changes on the affected and contralateral limb as assessed by skin thickness (Ultrasound).
Time Frame: Baseline and following a single treatment, an average of one hour
Measure: Mean (Full Range); unit: Percent Change
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Percent Change
  Affected Limb Percent Change | 116.1 [-46.5 to 310.3] | 5.6 [-17.0 to 76.1]
  Contralateral Limb Percent Change | 15.2 [-56.4 to 106.9] | 184.2 [-4.3 to 670.8]

5. Primary Outcome: Incidence of Adverse Events
Description: Adverse events reported between treatment and the 24-hour follow-up
Time Frame: 24-Hour Follow-Up
Measure: Count of Participants; unit: Participants
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

6. Primary Outcome: Post-Treatment Functional Vessel Assessment Via Near Infrared-fluorescent (NIRF) Imaging
Description: Comparison of the number of subjects with an increase in vessels for both the affected and contralateral limbs via near infrared-fluorescent (NIRF) imaging.
Time Frame: Baseline and following a single treatment, an average of one hour
Measure: Number; unit: Participants
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Participants
  Affected Limb | 0 | 0
  Contralateral Limb | 1 | 1

7. Primary Outcome: Projected Area or Extent of Dermal Backflow Via Near Infrared-fluorescent (NIRF) Imaging
Description: Comparison of the change in dermal backflow from the pre-treatment values to the post-treatment values as the sum of the volume of area for all locations for both the affected and contralateral limbs via near infrared-fluorescent (NIRF) imaging
Time Frame: Baseline and following a single treatment, an average of one hour
Measure: Number; unit: Percent Change
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Percent Change
  Affected Limb (Lateral Lower) | 65.4 | 20.6
  Contralateral Limb (Lateral Lower) | 0.0 | 0.0
  Affected Limb (Medial Lower) | 19.0 | -19.8
  Contralateral Limb (Medial Lower) | 0.0 | 0.0
  Affected Limb (Medial Upper) | 47.8 | 0.0
  Contralateral Limb (Medial Upper) | 0.0 | 0.0

8. Primary Outcome: Swelling in the Affected and Contralateral Limb as Assessed Using: Perometry (LymphaTech 3D Scanner)
Description: Compare the percent of participants by arm demonstrating a decrease in limb volume for the affected and contralateral limbs via Perometry (LymphaTech 3D Scanner)
Time Frame: Baseline and following a single treatment, an average of one hour
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Percentage of Participants
  Affected Limb | 0 | 100
  Contralateral Limb | 0 | 0

9. Primary Outcome: Skin Changes on the Affected and Contralateral Limb as Assessed by: Skin Thickness (Ultrasound)
Description: Comparison of the percent of participants by arm demonstrating a decrease in thickness for each site, separating skin and subcutaneous changes, on the affected limb via Ultrasound
Time Frame: Baseline and following a single treatment, an average of one hour
Measure: Number; unit: Percent of Participants
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
Percent of Participants
  Skin Thickness (Site A) | 100 | 100
  Skin Thickness (Site B) | 0 | 100
  Skin Thickness (Site C) | 0 | 100
  Subcutaneous Thickness (Site A) | 0 | 100
  Subcutaneous Thickness (Site B) | 0 | 0
  Subcutaneous Thickness (Site C) | 100 | 0

10. Primary Outcome: Absolute Change in Skin Thickness From Baseline to After Treatment
Description: Skin Changes on the affected and contralateral limb as assessed by skin thickness (Ultrasound).
Time Frame: Baseline and following a single treatment, an average of one hour.
Measure: Mean (Full Range); unit: mm
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
Number analyzed (Participants) | 1 | 1
mm
  Affected Limb Absolute Change | -1.70 [-8.25 to 0.11] | -0.03 [-1.18 to 0.6]
  Contralateral Limb Absolute Change | -0.52 [-1.86 to 0.31] | -1.54 [-6.44 to 0.04]

ADVERSE EVENTS:
Time Frame: Adverse event assessment will occur during the acute study period and ~24 hours after the acute study.
Arm/Group | Flexitouch Plus | Flexitouch Plus With SW
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04073823/Prot_SAP_000.pdf